CLINICAL TRIAL: NCT04493476
Title: Using a Herbal Remedy Extract for the Treatment of Endometriosis Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Yuval Kaufman, Dr yuval kaufman. Senior surgeon in the Department of Obstetrics and Gynecology, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0206-19COM2
Record Dates: First submitted 2020-07-07; First posted 2020-07-30 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2020-07

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: This is a prospective, placebo-controlled, double-blind randomized trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chineese Herbal formula (Active Comparator): The study group will be given capsules containing Chinese herbal formula extract - Traditional Chinese MedicinalSubstances
  Interventions: Drug: Chinese herbal formula
- placebo (Placebo Comparator): The control group tested will receive placebo capsules. Containing starch.
  Interventions: Drug: Chinese herbal formula

INTERVENTIONS:
Drug: Chinese herbal formula — Chinese herbal formula

SUMMARY:
A prospective, double-blind, placebo-controlled trial examining the effect of Chinese herbal medicine combined with curcumin defined as a dietary supplement on a study group of women with endometriosis, compared to control group.

research product:Chinese herbal extract and curcumin extract, which appear as nutritional supplements in the Ministry of Health database, the research product is packed in 800mg capsules.

Intended use: Composition of 14 different nutritional supplements, in Chinese herbal formula, for the treatment of endometriosis and its symptoms. The formula is formulated according to Chinese medicine principles and aims to reduce inflammation of the pelvic organs and reduce the levels of pain caused by endometriosis disease.

Objectives:Examine the Effect of Using Nutritional Supplements on Symptoms in Patients with Targeted Endometriosis Symptoms.

Primary Endpoints:

Benefit of pain in women suffering from symptoms of endometriosis patients taking herbal extract for 4 months of treatment.

Structure of the study:A prospective, double-blind, double-blind, placebo-controlled (randomized) placebo-controlled trial involving women suffering from endometriosis symptoms and meeting the inclusion and exclusion criteria and who agreed to participate in the study. The women will be randomly divided into the following two arms:

1. Study Group - Taking a daily dose of dietary supplement extract capsules
2. Control group - take a daily dose of Invo capsules Treatment efficacy will be measured according to a dedicated patient questionnaire with endometriosis symptoms that assess quality of life measures.

The study population will include 60 symptomatic women treated at the Multidisciplinary Center for Endometriosis Therapy at Lynn Medical Center.

DETAILED DESCRIPTION:
Endometriosis is a chronic and progressive gynecological disease, with an estimated invention of between 8-10% of women of childbearing age in the Western world . The disease is characterized by the presence of tissue resembling endometrial tissue . The tissue cells that are in the uterine space can settle on different organs in the pelvis. The cells continue to respond to the hormonal cycle as if they were inside the uterus and in each menstrual can grow and bleed. At the same time, an inflammatory process can be associated with various symptoms of pain. Symptoms are not specific but usually cyclical according to menstrual timing and include: severe menstrual cramps, heavy bleeding, diarrhea and constipation, infertility, urinary pain, recurrent infections, fainting, intercourse pain, leg pain and more.

The current practice is based on the removal of endometriosis lesions in surgery and / or drug therapy designed to suppress existing lesion activity and prevent lesion recurrence after surgery. To diagnose endometriosis in a definite way it is necessary to visually identify the lesions and by biopsy in surgery. In many patients, the symptoms of endometriosis can be treated pharmacologically and without surgery . Therefore, it is now widely accepted in many cases to treat pharmacologic anatomy empirically based on an estimated endometriosis-based diagnosis of appropriate anemia, gynecological examination, and vaginal ultrasound.

Very little has been investigated regarding the integration of endometriosis phenomena through complementary medicine that includes herbs and acupuncture, despite the vast clinical knowledge and experience gained. In the present study, we would like to examine the effect of complementary medicine that would include a combination of herbal remedies for pain symptoms in women with endometriosis.

In recent years, the Western world has begun to integrate complementary medicine in various treatments for chronic diseases and in particular endometriosis . The Chinese language review included 13 Chinese randomized clinical trials from 1994 to 2000. The studies included 1076 women who received Chinese herbs alone or in combination with recognized drugs . The proposed mechanism is that the herbs are involved in regulation of the endocrine and immune system and which improve blood flow and anti-inflammatory activity .

The ability of Chinese herbs to affect physiological changes indicates a mechanism of biological action of the herbs. However, the medicinal plants appear to have lower potency activity than synthetic drugs. They can contain an anti-inflammatory but less active ingredient than synthetic steroids.

Research Rationale Endometriosis is a chronic disease of infertile women. The main treatment is based on hormone drug therapy and surgical treatment. There are patients who, despite these treatments, still suffer from symptoms of endometriosis. There are also patients who are medically balanced but have to stop treatment for various reasons and need another non-hormonal response. Herbs have been found effective in treating gynecological problems and especially in chronic pelvic pain. They may relieve the symptoms in those women who wish to avoid hormone or surgical treatment or who are not symptomatically balanced despite the usual treatments.

The purpose of the study Investigate the effectiveness of treatment of symptoms and quality of life measures by the use of medicinal plants in women with symptoms of endometriosis.

Preliminary Results Primary Endpoints Benefit of pain indices in women suffering from symptoms of endometriosis between patients taking herbal extract and patients taking Invo for 4 months of treatment. Benefit is defined as a statistically significant improvement in VAS dimensions that will be examined by a daily journal and medical questionnaire.

Secondary Results Secondary Endpoints Quality-Of-Life Benefit Defined as a statistically significant improvement in questionnaire indices.

Also, a reduction in the use of painkillers and a lack of working days each month between the two groups.

The research product:Chinese herbal extract and curcumin extract, which appear as nutritional supplements in the Ministry of Health database, the research product is packed in 800mg capsules.

Intended use: Composition of 14 different nutritional supplements, in Chinese herbal formula, for the treatment of endometriosis and its symptoms. The formula is formulated according to Chinese medicine principles and aims to reduce inflammation of the pelvic organs and reduce the levels of pain caused by endometriosis disease.

Objectives:Examine the Effect of Using Nutritional Supplements on Symptoms in Patients with Targeted Endometriosis Symptoms.

Primary Endpoints:

Benefit of pain indices in women suffering from symptoms of endometriosis between patients taking herbal extract and patients taking Invo for 4 months of treatment.

Structure of the study:A prospective, double-blind, double-blind, placebo-controlled (randomized) placebo-controlled trial involving women suffering from endometriosis symptoms and meeting the inclusion and exclusion criteria and who agreed to participate in the study. The women will be randomly divided into the following two arms:

1. Study Group - Taking a daily dose of dietary supplement extract capsules
2. Control group - take a daily dose of Invo capsules Treatment efficacy will be measured according to a dedicated patient questionnaire with endometriosis symptoms that assess quality of life measures.

The study population will include 60 symptomatic women treated at the Multidisciplinary Center for Endometriosis Therapy at Lynn Medical Center.

ELIGIBILITY:
Inclusion Criteria:

1. Women with surgically diagnosed endometriosis and / or a clinical picture suitable for endometriosis.
2. Age 18 to 45. The patient is capable and willing to agree in writing ICF to enter the study.
3. There is no known allergy to any of the ingredients in the plant formula according to a sensitive patient's questioning.
4. The patient agrees to use contraception during the study period until the end of the medication if hormone therapy is not taken.
5. The patient has not changed / stopped / started hormone therapy in the previous three months of recruitment.

Exclusion Criteria:

Treated with kidney or liver disease, severe cardiovascular disease, chronic pancreatitis, diabetes or gallstones.

2. Treated with another cause of pain known. 3. Treated during pregnancy or breastfeeding. 4. A patient who is unable or unwilling to agree in writing for inclusion in the study.

5. Allergy is known to be one of the ingredients in the plant formula. 6. A patient who started hormone therapy, changed hormone therapy, or stopped in the three months prior to recruiting for the study.

7. Women who do not speak the Hebrew language about her ignorance

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 54 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Improvement in visual analogue scale pain scores in women with endometriosis symptoms treated with the herbal extract formula | 6 months
  Improvement will be measured by statistically significant visual analogue scale score differences collected by daily patient questionnaires

SECONDARY OUTCOMES:
Improvement in quality of life followiing treatment with the herbal extract formula | 6 months
  Statistically significant changes in QOL questionnaire scores and decrease in use of analgesics

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided